CLINICAL TRIAL: NCT06188741
Title: Phase 2 Trial of Selumetinib for the Prevention of Plexiform Neurofibroma Growth and Morbidity in Neurofibromatosis Type 1
Brief Title: Selumetinib for the Prevention of Plexiform Neurofibroma Growth in NF Type 1
Acronym: NF114
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Girish Dhall, MD, Chair of NFCTC, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010135; 164893 (Other: FDA - IND); W81XWH-22-3-0001 (Other Grant/Funding Number: DoD and Alexion)
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Intervention Model Description: Selumetinib (KoselugoTM) at the FDA approved dose of 25 mg/m2/dose PO BID
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: WBMRI for NF1 patients with no known PN (No Intervention): To assess the incidence of asymptomatic PN in any location in participants with NF1 and no known PN
- Part 2: Treatment randomization to selumetinib vs observation (Experimental): To determine if selumetinib treatment prevents PN growth in young participants with asymptomatic tumors in high-risk locations
  Interventions: Drug: Selumetinib
- Part 3: Part 2 participants with growing or symptomatic PN (Experimental): To assess the proportion of participants who are able to maintain tumor response after transition to an intermittent dosing schedule
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Selumetinib (KoselugoTM) at the FDA approved dose of 25 mg/m2/dose PO BID
  Other Names: Koselugo
  Arms: Part 2: Treatment randomization to selumetinib vs observation; Part 3: Part 2 participants with growing or symptomatic PN

SUMMARY:
Plexiform neurofibromas (PN) are known to cause significant morbidity in children with NF1. The recent FDA approval for selumetinib in children 2 years and older with inoperable symptomatic PN was based on the finding that selumetinib shrinks the majority of PN in children with NF1 and results in clinically meaningful benefit such as improvement in pain or range of motion. However, many morbidities, such as blindness or nerve damage, cannot be fully reversed with PN shrinkage. Therefore, there remains a critical need in this patient population to determine if young participants with PN in high-risk locations may benefit from early medical intervention prior to the development of clinical problems. This study will determine whether participants with asymptomatic PN in high-risk locations can potentially benefit from early treatment with selumetinib.

DETAILED DESCRIPTION:
Plexiform neurofibromas (PN) are known to cause significant morbidity in children with NF1. The recent FDA approval for selumetinib in children 2 years and older with inoperable symptomatic PN was based on the finding that selumetinib shrinks the majority of PN in children with NF1 and results in clinically meaningful benefit such as improvement in pain or range of motion. However, many morbidities, such as blindness or nerve damage, cannot be fully reversed with PN shrinkage. Therefore, there remains a critical need in this patient population to determine if young participants with PN in high-risk locations may benefit from early medical intervention prior to the development of clinical problems. This study will determine whether participants with asymptomatic PN in high-risk locations can potentially benefit from early treatment with selumetinib.

Other: This trial will be operated through the Neurofibromatosis Clinical Trials Consortium, funded by the Congressionally Directed Medical Research Program under the Department of Defense which consists of 24 sites throughout the United States.

Intervention: Selumetinib (KoselugoTM) at the FDA approved dose of 25 mg/m2/dose PO BID.

Study Duration: 7 years Partcipant Durations: 5 years

ELIGIBILITY:
PART 1:

Inclusion Criteria:

1. Age: > 1 (>12 months) and ≤8 years of age at the time of study enrollment.
2. Diagnosis: Participants with a diagnosis of NF1 based on the 2021 revised consensus criteria [52] and
3. No known PN (prior to enrollment on Part 1). Participants for whom there is clinical suspicion for a PN (e.g., subtle facial asymmetry or large overlying hyperpigmented area) may be included in the study after discussion with the Study Chair so long as they have not previously had an MRI of the region of concern and are otherwise asymptomatic.
4. Physical exam at your institution within 1 year prior to consent.
5. Written informed consent must be obtained from the legal guardians of all participants <18 years of age.

Exclusion Criteria:

1. Presence of a known, symptomatic PN with or without previous MRI imaging.
2. Patients who have had previous whole-body MRI (WBMRI) are excluded from the study. However, patients who have had regional MRI(s) for an indication other than a PN and did not have a PN identified on previous MRI may still be eligible for the study.
3. Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol.
4. Prior treatment with selumetinib or another specific MEK1/2 inhibitor.
5. Evidence of an optic pathway or other low-grade glioma, high grade glioma, malignant peripheral nerve sheath tumor, or other cancer/tumor requiring treatment with chemotherapy, biologic therapy or radiation therapy.
6. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at a tumor, immunotherapy, or biologic therapy.
7. Clinical judgement by the investigator that the patient should not participate in the study.

PART 2:

Inclusion Criteria:

1. Enrolled on Part 1 of this study and completed baseline WBMRI within 6 weeks of planned enrollment on Part 2.
2. A measurable (≥3 mL) PN in a high-risk location as defined below (this must be confirmed by Study Chair or a member of the Study Committee prior to enrollment on Part 2).

   * In the head or neck (with the exception of isolated scalp lesions) OR
   * Within the brachial or lumbosacral plexus OR
   * Adjacent to high-risk structure(s), defined as:

     1. Major ("named") blood vessel OR
     2. Major ("named") airway OR
     3. Hollow viscus OR
     4. Spinal cord and foramina OR
     5. Vital Organs (including heart, lungs, liver, spleen, etc.)
3. Body Surface Area (BSA): BSA ≥ 0.55 m2 [pending availability of granule formulation].
4. Performance status: Lansky performance ≥70%. Participants who are wheelchair bound because of paralysis or immobility secondary to a non-PN related manifestation of NF1 (such as tibial pseudarthrosis or severe scoliosis) should be considered ambulatory when they are in their wheelchair.
5. Able to swallow whole capsules [Pending availability of granule formulation].
6. Hematologic Function: Absolute neutrophil count ≥1200/µL, hemoglobin ≥9g/dL, and platelets ≥100,000/µL (without transfusions).
7. Hepatic Function: Bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within ≤ 3 x upper limit of normal.
8. Renal Function: Creatinine clearance or radioisotope GFR ≥60ml/min/1.73 m2 or a normal serum creatinine based on age, described in the table below.

   Age (years) Maximum Serum Creatinine (mg/dL)

   ≤5 0.8 >5 to ≤10 1.0 >10 to ≤15 1.2 >15 1.5
9. Cardiac Function:

   1. Normal ejection fraction (ECHO or cardiac MRI) ≥ 53% (or the institutional normal; if a range is given then the upper value of the range will be used).
   2. EKG with QTC or QTcF ≤450 msec.
10. Adequate Blood Pressure defined as:

    A blood pressure (BP) ≤ the 95th percentile for age, height, and gender. Adequate blood pressure can be achieved using medication for treatment of hypertension. Participants must be on stable antihypertensive regimen for at least 30 days prior to study entry.
11. Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
12. Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g., grapefruit juice or marmalade) during the study, as these may affect selumetinib metabolism.

Exclusion Criteria:

1. Evidence of an optic pathway or other low-grade glioma, high-grade glioma, malignant peripheral nerve sheath tumor, or other cancer/tumor requiring treatment with chemotherapy, biologic therapy or radiation therapy.
2. Ongoing radiation therapy, chemotherapy, hormonal therapy, immunotherapy, or biologic therapy directed at a tumor.
3. Prosthesis, orthopedic implant, or dental braces that would interfere with volumetric analysis of target PN on MRI.
4. Use of an investigational agent within the past 30 days.
5. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses, or renal transplant, including any patient known to have hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) will be excluded.
6. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
7. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
8. Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to initiation of therapy.
9. Participants not achieving adequate blood pressure despite antihypertensive therapy for control of blood pressure.
10. Cardiac conditions:

    1. Known inherited coronary disease
    2. Symptomatic heart failure (NYHA Class II-IV prior or current cardiomyopathy, or severe valvular heart disease)
    3. Prior or current cardiomyopathy
    4. Severe valvular heart disease
    5. History of atrial fibrillation
11. Ophthalmologic conditions:

    1. Current or past history of central serous retinopathy or retinal pigment epithelial detachment (RPED).
    2. Current or past history of retinal vein occlusion.
    3. History of radiation therapy that included the orbit in the field of treatment.
    4. Known intraocular pressure (IOP) > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Participants with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the Study Chair.
    5. Participants with any other significant abnormality on ophthalmic examination should be discussed with the Study Chair for potential eligibility.
    6. Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) will NOT be considered a significant abnormality for the purposes of the study.
12. Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib.
13. Recent major surgery within a minimum of 4 weeks prior to starting study treatment.
14. Any unresolved chronic toxicity with CTCAE grade ≥ 2 from previous therapy, except for alopecia.
15. Receiving herbal supplements or medications known to be strong or moderate inhibitors or inducers of the cytochrome P450 (CYP)2C19 and CYP3A4 enzymes or fluconazole unless such products can be safely discontinued at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication.

PART 3:

Inclusion Criteria:

1. Enrolled on Part 2 of this study and had PN growth >20% OR development of PN related symptom(s) while on observation portion of Part 2 (including the first 2 years for the observation arm OR during first year of observation after treatment with selumetinib).
2. Body Surface Area (BSA): BSA ≥ 0.55 m2 [pending availability of granule formulation].
3. Performance status: Lansky performance ≥70%. Participants who are wheelchair bound because of paralysis or immobility secondary to a non-PN related manifestation of NF1 (such as tibial pseudarthrosis or severe scoliosis) should be considered ambulatory when they are in their wheelchair.
4. Able to swallow whole capsules [Pending availability of granule formulation].
5. Hematologic Function: Absolute neutrophil count ≥1200/µL, hemoglobin ≥9g/dL, and platelets ≥100,000/µL (without transfusions).
6. Hepatic Function: Bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within ≤ 3 x upper limit of normal.
7. Renal Function: Creatinine clearance or radioisotope GFR ≥60mL/min/1.73 m2 or a normal serum creatinine based on age, described in the table below.

   Age (years) Maximum Serum Creatinine (mg/dL)

   ≤5 0.8 >5 to ≤10 1.0 >10 to ≤15 1.2 >15 1.5
8. Cardiac Function:

   1. Normal ejection fraction (ECHO or cardiac MRI) ≥ 53% (or the institutional normal; if a range is given then the upper value of the range will be used).
   2. EKG with QTC or QTcF ≤450 msec.
9. Adequate Blood Pressure defined as:

   A blood pressure (BP) ≤ the 95th percentile for age, height, and gender. Adequate blood pressure can be achieved using medication for treatment of hypertension. Participants must be on stable antihypertensive regimen for at least 30 days prior to study entry.
10. Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
11. Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g., grapefruit juice or marmalade) during the study, as these may affect selumetinib metabolism.

Exclusion Criteria:

1. Evidence of an optic pathway or other low-grade glioma, high-grade glioma, malignant peripheral nerve sheath tumor, or other cancer/tumor requiring treatment with chemotherapy, biologic therapy or radiation therapy.
2. Ongoing radiation therapy, chemotherapy, hormonal therapy, immunotherapy, or biologic therapy directed at a tumor.
3. Prosthesis, orthopedic implant, or dental braces that would interfere with volumetric analysis of target PN on MRI.
4. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses, or renal transplant, including any patient known to have hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) will be excluded.
5. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
6. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
7. Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to initiation of therapy.
8. Participants not achieving adequate blood pressure despite antihypertensive therapy for control of blood pressure.
9. Cardiac conditions:

   1. Known inherited coronary disease
   2. Symptomatic heart failure (NYHA Class II-IV prior or current cardiomyopathy, or severe valvular heart disease)
   3. Prior or current cardiomyopathy
   4. Severe valvular heart disease
   5. History of atrial fibrillation
10. Ophthalmologic conditions:

    1. Current or past history of central serous retinopathy or retinal pigment epithelial detachment (RPED).
    2. Current or past history of retinal vein occlusion.
    3. History of radiation therapy that included the orbit in the field of treatment.
    4. Known intraocular pressure (IOP) > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Participants with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the study chair.
    5. Participants with any other significant abnormality on ophthalmic examination should be discussed with the Study Chair for potential eligibility.
    6. Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) will NOT be considered a significant abnormality for the purposes of the study.
11. Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib.
12. Recent major surgery within a minimum of 4 weeks prior to starting study treatment.
13. Any unresolved chronic toxicity with CTC AE grade ≥ 2 from previous therapy, except for alopecia.
14. Receiving herbal supplements or medications known to be strong or moderate inhibitors or inducers of the cytochrome P450 (CYP)2C19 and CYP3A4 enzymes or fluconazole unless such products can be safely discontinued at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 60 months
  Progression free survival (PFS) in the group treated with selumetinib compared to those in the observation group

SECONDARY OUTCOMES:
Participants found to have a previously unknown measurable PN | 60 months
  Proportion of participants found to have a previously unknown measurable PN in any location on WBMRI imaging
PFS | 60 months
  2) PFS through one year after transitioning from continuous to an intermittent dosing schedule

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Childrens of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children/Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Cancer Institute/ National Institutes of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No